CLINICAL TRIAL: NCT03535220
Title: The American Society of Hematology (ASH) Research Registry: A Multicenter Research Registry of Patients With Hematologic Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: American Society of Hematology (Other)
Responsible Party: Sponsor
Other Study IDs: 1185686
Record Dates: First submitted 2018-05-11; First posted 2018-05-24 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Benign and Malignant Hematologic Diseases
Keywords: Multiple Myeloma; Sickle Cell Disease
MeSH Terms: conditions — Multiple Myeloma; Anemia, Sickle Cell | interventions — Protease Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Observational/ Interventional: Hematologic Disease
  Interventions: Combination Product: Protease Inhibitors

INTERVENTIONS:
Combination Product: Protease Inhibitors — Nucleic Acid Synthesis Inhibitors,Hydroxyurea,Antineoplastic Agents
  Other Names: Monoclonal Antibodies Proteasome inhibitors,

SUMMARY:
This is a multicenter, retrospective and prospective, long-term registry of patients with benign or malignant hematologic diseases, whether or not these patients were or were not treated with disease-specific treatments. Information will be collected on patient demographics, disease characteristics, genomic and molecular data, laboratory data, pathology, radiographic reports, clinical status, quality of life, medications, and dosing information. Where appropriate, these data structures may be based on a combination of Fast Healthcare Interoperability Resources (FHIR) , Consolidated-Clinical Data Architecture (C-CDA) and/or client-speciﬁc structure deﬁnitions.

DETAILED DESCRIPTION:
The primary goal of the ASH Registry is to further the scientific knowledge base for the diagnosis, understanding, and management of benign and malignant hematologic conditions by assembling data collected in usual care and clinical trials. Secondary goals are to characterize and study practice patterns for benign and malignant hematologic conditions in usual clinical practice, and to aggregate patient-reported data to further understand and improve the patient experiences of those affected by these conditions. These objectives will be fulfilled by amassing previously collected data within institutions and networks, and by building consortia of institutions and networks to support prospective data collection efforts.

As a research-focused effort, another objective of the ASH Registry is to create a learning community of hematologic researchers and clinicians by inviting collaborative analyses and publications of the data that are collected within it. These analyses may be valuable to basic and translational researchers developing new lines of scientific inquiry; clinical researchers studying the safety and efficacy of hematologic therapies in current practice; industry participants developing new therapies or new indications for previously developed treatments; regulators who are interested in new endpoints and other insights to facilitate the evaluation of novel approaches; and patients who are looking to understand how hematologic diseases and treatments for these diseases will affect their lives. As these different stakeholder groups come together to develop and disseminate these analyses, the ASH Registry will further expand to accommodate additional data collection to address yet unanswered questions that follow.

ELIGIBILITY:
Inclusion Criteria:

* Patients (>18 years of age) must have diagnostically- or investigator-confirmed benign or malignant hematologic disease.
* For prospective data collection efforts within the ASH Registry that require informed consent, children (<18 years of age) with hematologic disease whose parent/legal guardian consents on their behalf may be included.

Exclusion Criteria:

* Adults that are unable to consent.
* Prisoners

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and Adult population
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2018-05-10 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Minimal Residual Disease | Up to 5 Years
  Cancer cells from the bone marrow) that remain in the patient during treatment, or after treatment when the patient is in remission e.g. 3 months, 6 months, one year, or end of current treatment.

SECONDARY OUTCOMES:
Patient reported outcomes (health-related QoL ) | Up to 5 Years
  Health-related QoL

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Thompson, MD,MPH, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- American Society of Hematology, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided